CLINICAL TRIAL: NCT01002495
Title: A Phase I/II Open Label, Dose-Escalation Study to Assess the Safety and Tolerability of VM202 in Subjects With Chronic Refractory Myocardial Ischemia
Brief Title: Gene Therapy for the Treatment of Chronic Stable Angina
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was never initiated at any sites.
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMCAD-001/B
Record Dates: First submitted 2009-10-24; First posted 2009-10-27 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Ischemia
Keywords: myocardial; ischemia; coronary disease; angina
MeSH Terms: conditions — Myocardial Ischemia; Ischemia; Coronary Disease; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Eight endocardial injection for a total dose of 1mg VM202
  Interventions: Biological: VM202
- Cohort 2 (Experimental): Eight endocardial injections for a total dose of 2mg VM202
  Interventions: Biological: VM202
- Cohort 3 (Experimental): Twelve endocardial injections for a total dose of 3mg VM202
  Interventions: Biological: VM202

INTERVENTIONS:
Biological: VM202 — Endocardial injections on Day 0.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of catheter based injections of VM202 into the heart.

DETAILED DESCRIPTION:
A phase I/II, open label, dose-escalation, multicenter, 12 month study designed to assess the safety and tolerability of catheter based percutaneous myocardial injection of VM202 in patients with chronic refractory myocardial ischemia. The study will consist of three (3) cohorts with a total of 4 subjects enrolled in each cohort. Endocardial injections will be performed with the MyoStar Injection Catheter under guidance of the NOGA XP Cardiac Navigation System.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years, but less than or equal to 75 years.
* Stable chronic refractory angina classified as Canadian Cardiovascular Society (CCS) functional class II - IV
* Left ventricular ejection fraction (LVEF) of ≥30% and ≤ 50%;
* Clinical signs and symptoms of significant ischemia by treadmill test or Stress imaging (SPECT, Echo or CARDIAC MRI acceptable)
* Subjects must be able to complete a minimum of 3 minutes, but no more than 10 minutes on a Modified Bruce treadmill protocol.
* Patients on maximal medical therapy including at least 2 of the following (unless hemodynamic parameters or intolerance contraindicate their use):(a) Long acting nitrate, (b) Beta Blocker or (c) Calcium Channel Blocker (d) Ranolazine. Optimal medical regimen for each subject will be decided by the referring cardiologist or principal investigator. Patients must be on stable medical regimen for 30 days prior to enrollment.
* Coronary angiogram within 1 year to confirm the presence of coronary disease which is not amenable to standard revascularization procedures.
* Candidates must not be eligible for any other revascularization procedures. The participant and his/her coronary film must have been discussed with an independent cardiac surgeon and must have been denied for CABG or PTCA. Participants who are marginal or poor candidates for conventional revascularization will be considered eligible if the risks of performing a CABG or PTCA procedure outweigh the potential benefit and/or such a procedure is unlikely to offer a worthwhile clinical benefit. The criteria defining such cases may include, but may not be limited to, the following examples:

  * Diffuse or distal vessel disease
  * Chronic occlusions
  * Unprotected left main stenosis
  * Tortuous or severely angulated vessels
  * Severely calcified vessels
  * Small vessels (< 2.5mm)
* Subjects with childbearing potential must take acceptable measure to prevent pregnancy during the course of the study.
* Subject capable of understanding with the protocol and signing the informed consent document prior to any study related procedure.

Exclusion Criteria:

* Subjects who have undergone a successful revascularization procedure within 6 months of enrollment;
* MI, unstable angina requiring > 24 hour hospitalization, or percutaneous coronary intervention, within last 90 days;
* Stroke or TIA within last 180 days;
* Predominant CHF symptoms;
* Hemodynamically significant severe primary valvular heart disease, unless corrected by a properly functional prosthetic valve;
* Uncontrolled hypertension as defined as systolic BP 170 mmHg or diastolic > 90 mmHg at baseline/ screening evaluation;
* Sustained ventricular tachycardia or automatic implantable cardiodefibrillator (AICD) firing within last 180 days;
* History of ventricular fibrillation;
* Use of the MyoStar catheter may not be appropriate for patients with prosthetic valves. Patients with a mechanical valve at risk for injury due to the interventional approach should be excluded;
* Subjects with any comorbidity that may interfere with the ability to perform a maximal treadmill test (e.g. severe arthritis, musculoskeletal disorders, COPD);
* Subjects with a history of malignancy, a known active malignancy, or a new screening finding of malignant neoplasm;
* Patients with family history of colon cancer in any first degree relative unless they have undergone a colonoscopy in the last 12 months with negative findings;
* Elevated PSA unless prostate cancer has been excluded;
* Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination.

  * Cataract surgery within 6 months of trial;
  * Vascular lesions of the anterior segment of the eye (infection or ulceration of the cornea, rubeotic glaucoma, etc);
  * Vascular lesions of the posterior segment of the eye or proliferative retinopathy in diabetics, macular edema, s/p photocoagulation for macular edema or proliferative retinopathy; nondiabetics with central or branch retinal vascular occlusions, sickle cell retinopathy, ischemic retinopathy due to retinal venous stasis or carotid artery disease);
  * Choroidal new vessels associated with age-related macular degeneration, myopic degeneration, presumed ocular histoplasmosis syndrome, angioid streaks, pseudoxanthoma elasticum, or without ocular disease; and
  * Large elevated choroidal nevi, choroidal vascular tumors (choroidal hemangioma), or melanomas.
* Chronic inflammatory disease (e.g. Crohn, Rheumatoid Arthritis);
* Active infectious disease and/or known to have tested positive for human immunodeficiency virus (HIV), human t lymphotrophic virus (HTLV), hepatitis B virus (HBV), or hepatitis C virus (HCV);
* Specific laboratory values at Screening including: Hemoglobin < 9.0, g/dL, WBC < 3,000 cells per microliter, platelet count <75,000/mm3, Creatinine > 2.0 mg/dL, AST and/or ALT > 3 times the upper limit of normal or any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary;
* Patients have undergone enhanced external pulsation (EECP) treatment within the last 6 months;
* Pregnancy or lactation;
* Severe comorbidity associated with a reduction of life expectancy of less than 1 year;
* Exposure to any previous experimental angiogenic therapy and/or myocardial laser therapy; or therapy with another investigational drug within 180 days of enrollment or participation in any concurrent study that may confound the results of this study;
* Major psychiatric disorder in past 6 months;
* History of recent tobacco abuse (within past < 5 years);
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Estimated); Primary Completion 2015-07 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The primary study objective is to evaluate safety and tolerability of a catheter-based, endocardial injection of different doses of VM202. | Days 1, 7, 14, 21, 30, 60, and 90, 6 and 12 months

SECONDARY OUTCOMES:
Secondary objectives include the assessment of the angiogenic potential of VM202 | one month, three months, six months and twelve months
Efficacy measures include exercise treadmill test, SPECT, cardiac MRI and change in use of anti-anginal medications. | Days 1, 7, 14, 21, 30, 60, and 90. 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Minneapolis Heart Institute Foundation/ Abbott Northwestern Hospital, Minneapolis, Minnesota